CLINICAL TRIAL: NCT05824819
Title: "Is the Reduced Quality of Life of Women With Endometriosis the Result of Peritoneal Dysbiosis?"
Brief Title: Endometriosis and Peritoneal Dysbiosis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jagiellonian University (Other)
Responsible Party: Principal Investigator, Iwona Magdalena Gawron, Ph.D., Principal Investigator, Jagiellonian University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 1072.6120.24.2023
Record Dates: First submitted 2023-03-22; First posted 2023-04-24 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Endometriosis; Infertility Unexplained
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Intervention Model Description: Prospective tertiary single-centre cohort study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Endometriosis (Active Comparator): Women subjected to laparoscopy due to endometriosis. Before the procedure: collection of a stool sample for NGS testing (2 ml); During the procedure: collection of fluid/ washings from the peritoneal cavity (2 ml) and fluid from the endometrial cyst (2 ml), and collection of endometrial tissue by aspiration biopsy of the uterine cavity (1 ml) for NGS examination.
  Interventions: Diagnostic Test: Next Generation Sequencing (NGS)
- Idiopathic infertility (Active Comparator): Women subjected to laparoscopy due to idiopathic infertility. Before the procedure: collection of a stool sample for NGS testing (2 ml); During the procedure: collection of fluid/ washings from the peritoneal cavity (2 ml) and collection of endometrial tissue by aspiration biopsy of the uterine cavity (1 ml) for NGS examination.
  Interventions: Diagnostic Test: Next Generation Sequencing (NGS)

INTERVENTIONS:
Diagnostic Test: Next Generation Sequencing (NGS) — Biological materials (stool, peritoneal/ovarian cyst fluid, endometrial aspirate) will be secured and then subjected to molecular analysis using the Next Generation Sequencing (NGS) method. The stages will include: i) isolation of bacterial DNA from biological materials, ii) preparation of libraries for sequencing, including the performance of the PCR and nested-PCR methods on bacterial DNA isolates from the tested samples of biological materials, iii) purification of amplification products, indexing, validation of the concentration of amplicons, pooling and denaturation of libraries, iv) standardization and optimization of the procedure for the isolation of bacterial metagenomic DNA from biological materials from intestines, peritoneal cavity, uterine cavity and endometrial tissues, v) standardization of the nested-PCR method on bacterial DNA isolates from the tested biological materials, vi) submission of samples for sequencing.

SUMMARY:
Endometriosis is a complex clinical syndrome that impairs many aspects of a woman's life, characterized by a chronic estrogen-dependent inflammatory process, mainly affecting the pelvic organs, with ectopic presence of tissue analogous to the uterine mucosa (endometrium). Despite intensive research in the field of etiopathogenesis, its cause has not yet been determined, and treatment remains symptomatic. Endometriosis causes two main complications, i.e. pelvic pain syndrome and infertility. In recent years, thanks to the analysis of the human microbiome, it has become possible to deepen the knowledge of the physiological and pathological interactions between microorganisms inhabiting various body areas and the host. Bacteria may enter the peritoneal cavity in the mechanism of retrograde menstruation and translocate from the intestines, and then promote the development of local and systemic inflammation, leading to the symptoms of endometriosis. The study is to determine whether the presence of a specific intestinal, peritoneal and uterine microbiome correlates with endometriosis stage and whether its presence predisposes to increased pain or infertility. Concordance or divergence of bacterial populations inhabiting the peritoneal and uterine cavities could have clinical implications, i.e. the possibility of empirical antibiotic therapy in patients undergoing only endometrial aspiration biopsy and not opting for surgical treatment.

DETAILED DESCRIPTION:
The main objective of the project is to analyze gut, peritoneal and uterine microbiome in women who undergo laparoscopy due to endometriosis (arm 1) or idiopathic infertility (arm 2). Detailed objectives are: i) analysis of the correlation between the composition of the intestinal, peritoneal and uterine microbiome with the stage of endometriosis according to ASRM, ii) qualitative comparison of the intestinal and peritoneal microbiome to the uterine cavity microbiome in women with endometriosis vs. idiopathic infertility, iii) analysis of the correlation between the composition of the intestinal, peritoneal and uterine microbiome with the intensity of pain and infertility, iv) comparing the quality of life in both arms and assessing its correlation with the local microbiome. Quality of life will be assessed in both arms using the SF-36 questionnaire, and then compared. The SF-36 self-reported questionnaire covers eight health domains: physical functioning (10 items), bodily pain (2 items), role limitations due to physical health problems (4 items), role limitations due to personal or emotional problems (4 items), emotional well-being (5 items), social functioning (2 items), energy/fatigue (4 items), and general health perceptions (5 items). Scores for each domain range from 0 to 100, with a higher score defining a more favorable health state. The study group will consist of women of childbearing age, undergoing surgical treatment due to pelvic endometriosis or idiopathic infertility. Before the surgery, a stool sample will be taken for examination of intestinal microbiome. During scheduled laparoscopy, in addition to the planned procedure, which is the purpose of hospitalization, an endometrial aspiration biopsy will be performed and fluid from the peritoneal cavity and/or fluid from the ovarian cyst will be collected for analysis of the local microbiome. Biological materials (stool, peritoneal/ovarian cyst fluid, endometrial aspirate) will be secured and then subjected to molecular analysis using the Next Generation Sequencing (NGS) method. The stages will include: i) isolation of bacterial DNA from biological materials, ii) preparation of libraries for sequencing, including the performance of the PCR and nested-PCR methods on bacterial DNA isolates from the tested samples of biological materials, iii) purification of amplification products, indexing, validation of the concentration of amplicons, pooling and denaturation of libraries, iv) standardization and optimization of the procedure for the isolation of bacterial metagenomic DNA from biological materials from intestines, peritoneal cavity, uterine cavity and endometrial tissues, v) standardization of the nested-PCR method on bacterial DNA isolates from the tested biological materials, vi) submission of samples for sequencing. Sequencing data will be subjected to bioinformatics analysis to obtain bacterial profiles (the percentage composition of the local bacterial population by phyla and genera). The aim is to characterize the microbiome of the intestines, peritoneal and the uterine cavity in women undergoing surgical treatment for endometriosis or invasive diagnostics for idiopathic infertility, and to compare the bacterial populations in these locations, which may also provide information on the origin of bacteria in the peritoneal cavity.

ELIGIBILITY:
Inclusion Criteria:

* age 18-45 years
* indications for surgical treatment of endometriosis by laparoscopy and/or indications for invasive diagnostics by laparoscopy due to idiopathic infertility.

Exclusion Criteria:

* abdominal surgeries performed within 6 months prior hospitalisation
* active infection of the genital tract
* inflammatory bowel disease
* antibiotic therapy and use of probiotics within 3 months before surgery

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Composition of intestinal, peritoneal and uterine microbiome in both study arms | up to 6 months
  Percentage composition of the local bacterial population by phyla and genera

SECONDARY OUTCOMES:
Relation of the composition of intestinal, peritoneal and uterine microbiome and endometriosis stage | up to 6 months
  Correlation between the percentage composition of the local bacterial population (by phyla and genera) and the ASRM endometriosis stage
Relation of the uterine microbiome to the intestinal and peritoneal microbiome in women with endometriosis and idiopathic infertility | up to 6 moths
  Correlation between the percentage composition of the uterine bacterial population (by phyla and genera) and the percentage composition of the intestinal and peritoneal microbiome (by phyla and genera)
Relation of intestinal, peritoneal and uterine microbiome and symptoms | up to 6 moths
  Correlation between the percentage composition of local microbiomes (by phyla and genera) and the severity of pain symptoms on the Numeric Rating Scale (NRS from 0 - no pain to 10 - maximum pain) and the duration of infertility (in years)
Composition of intestinal, peritoneal and uterineand quality of life | up to 6 moths
  Correlation between the percentage composition of local microbiomes (by phyla and genera) and the percentage result of the SF-36 questionnaire evaluating of 8 area of life on a scale from 0% - the worst quality to 100% - the best quality

CONTACTS AND LOCATIONS:
Overall Officials: Robert Jach, Prof. Ph.D., Study Chair — Jagiellonian University
Locations (1):
- Jagiellonian University Medical College, Department of Gynecology and Obstetrics, Krakow, Poland

IPD SHARING:
Plan to Share IPD: No